CLINICAL TRIAL: NCT03037983
Title: Improving Neurocognitive Deficits and Function in Schizophrenia With Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Stanford University (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: D2382-P; 12246865 (Other Grant/Funding Number: Veterans Affairs - Rehabilitation R&D); 38101 (Other: Stanford IRB)
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Transcranial magnetic stimulation; Electroencephalography
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Subjects will receive actual rTMS treatment.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham rTMS (Sham Comparator): Subjects will attend and sit through the session, but no rTMS treatment will be actually delivered to them.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — rTMS is a non-invasive procedure, in which the administration of a transient magnetic field induces electrical currents in specific, targeted brain regions. The intervention will be administered in 20 sessions lasting 50 minutes each over the course of 2-6 weeks. Up to two sessions may be scheduled per day with a one-hour interval in-between.
  Other Names: rTMS
  Arms: Active rTMS
Device: Sham — Subjects will still attend treatment sessions as outlined in the rTMS intervention. However, the device will not deliver any stimulation to the subject.
  Arms: Sham rTMS

SUMMARY:
The purpose of this study is to determine whether repetitive transcranial magnetic stimulation (rTMS) is effective in remediating cognitive deficits while also improving functionality in Veterans with schizophrenia.

DETAILED DESCRIPTION:
High-frequency, repetitive transcranial magnetic stimulation (rTMS) to the dorsolateral prefrontal cortex (DLPFC), the dysfunctional brain region most implicated in cognitive deficits in schizophrenia, has recently been shown to improve cognition in non-Veteran samples with schizophrenia. The investigators' goal is to confirm the efficacy of this treatment modality to remediate cognitive deficits and improve functionality in Veterans with schizophrenia, as well as to gain a better understanding of the neural mechanisms responsible for cognitive deficits and their remediation. The investigators propose conducting a small-scale study to generate pilot data supporting the feasibility of conducting rTMS with Veterans and the effectiveness of rTMS in this population. In addition, the investigators will conduct neurophysiologic experiments to test whether certain neural maker of abnormal brain function improves with rTMS.

ELIGIBILITY:
Inclusion Criteria:

* SCID (Structured Clinical Interview for DSM Disorders) confirmed diagnosis of Schizophrenia or Schizoaffective Disorder
* Stable medication regimen (no change in dose or agents within the 2 weeks prior to study entry and throughout the duration of the study)
* Stable social environment and housing to enable regular attendance at clinic visits
* Ability to undergo cognitive testing, EEG scans and rTMS
* IQ (intelligence quotient) > 80 (WASI full scale score)
* In general good medical health
* Is in treatment with a psychiatrist and/or primary care physician within the VHA (Veteran's Health Administration) system

Exclusion Criteria:

* Pregnant or lactating female
* History of prior adverse reaction to TMS
* On medications known to significantly lower seizure threshold, e.g.:

  * clozapine
  * chlorpromazine
  * clomipramine
* History of seizures or conditions known to substantially increase risk for seizures
* Implants or medical devices incompatible with TMS
* Acute or unstable chronic illness that would affect participation or compliance with study procedures, e.g.:

  * unstable angina
* Substance abuse/dependence (not including caffeine or nicotine) within one-month period prior to study entry or during study participation
* Unstable psychiatric symptoms that precludes consistent participation in the study, e.g.:

  * active current suicidal intent or plan
  * severe psychosis
* History of loss of consciousness greater than 15 minutes due to head injury.
* Participation in another concurrent clinical trial
* Patients with prior exposure to rTMS
* Have a mass lesion, cerebral infarct or other active central nervous system disease, or history of traumatic brain injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong H. Yoon, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the approached potential participants, many were unable to participate due to difficulties with the amount of time required to participate in the study, or a change in interest.
Groups:
- Active: Subjects will receive actual rTMS treatment.
  Repetitive transcranial magnetic stimulation: rTMS is a non-invasive procedure, in which the administration of a transient magnetic field induces electrical currents in specific, targeted brain regions. The intervention will be administered in 20 sessions lasting 50 minutes each over the course of 2-6 weeks. Up to two sessions may be scheduled per day with a one-hour interval in-between.
- Sham: Subjects will attend and sit through the session, but no rTMS treatment will be actually delivered to them.
  Sham: Subjects will still attend treatment sessions as outlined in the rTMS intervention. However, the device will not deliver any stimulation to the subject.
Period: Overall Study
Arm/Group | Active | Sham
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.2) | 40.5 (14.5) | 45.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
Brief Assessment of Cognition in Schizophrenia (BACS) Composite T-score Score at Baseline [Mean (Standard Deviation); unit: T-score] — The Brief Assessment of Cognition in Schizophrenia (BACS) represents cognitive ability of people with schizophrenia, where scores from six sub-scales of cognition were normalized to a composite T-score in which the normalized T-score has a mean of 50 and S.D. of 10 of the reference groups, where a higher score significantly above the mean indicates greater cognitive ability. Alternatively, scoring significantly below the mean would indicate lower cognitive ability as reflected in the data.
  T-score | 33.75 (10.10) | 33.5 (10.66) | 33.62 (10.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Working Memory Function
Description: Changes in scores for working memory performance accuracy will serve as dependent measure for testing the hypothesis that rTMS improves working memory. Working memory performance was assessed using a non-standardized task developed in house, which is basically a Sterberg style delayed response task in which memoranda are displayed and are to be remembered across a short delay period. The hypothesis will be supported if the investigators find greater working memory difference in the active compared to the sham-rTMS-treated groups as revealed by t-tests and two-sided tests at an alpha level of 0.05. Scores will be reported as a change in percent accuracy during this working memory task, where higher percent accuracy is better and scores range from -100% to 100%.
Time Frame: before treatment and after 6-week treatment
Measure: Mean (Standard Deviation); unit: % change in Working Memory Task Accuracy
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 4
% change in Working Memory Task Accuracy | -7.28 (12.95577091) | -5.9 (15.55040192)
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = .849, t-test, 2 sided; Mean Difference (Net) = 1.38

2. Primary Outcome: Change in Neurophysiologic Function
Description: Gamma oscillation is viewed as a measure of neurophysiologic function. The investigators will be conducting task-evoked electroencephalography (EEG) to measure gamma oscillation before and after rTMS. It is predicted that the intervention will improve gamma oscillations.
Time Frame: before treatment and after 6-week treatment
Measure: Mean (Standard Deviation); unit: wavelet coefficient in dB
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 4
wavelet coefficient in dB | 0 (.025) | 0 (.03)

3. Primary Outcome: Change in Level of Everyday Functioning
Description: Changes in Global Functioning Scale scores (GF) will serve as dependent measure for testing the hypothesis that rTMS improves functioning. The hypothesis will be supported if the investigators find greater GF-difference in the active compared to the sham-rTMS-treated groups as revealed by t-tests and two-sided tests at an alpha level of 0.05.
  Scale's values range from a minimum score of 1 to a maximum score of 10, with a higher score means better functioning.
Time Frame: before treatment and after 6-week treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 4
score on a scale | 0 (3.1) | -.5 (1.7)
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = .782, t-test, 2 sided — t = 0.287; Mean Difference (Net) = 0.5

4. Primary Outcome: Change in General Cognitive Ability
Description: Changes in Brief Assessment of Cognition (BACS) score will serve as a dependent measure for testing the hypothesis that rTMS improves cognitive functioning. The hypothesis will be supported if the investigators find greater GF-difference in the active compared to the sham-rTMS-treated groups as revealed by t-tests and two-sided tests at an alpha level of 0.05. Data will be reported as change in Z-score on the scale, where a higher value means a better outcome, with scores ranging from -3 to 3.
Time Frame: before treatment and after 6-week treatment
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Sham
Number analyzed (Participants) | 5 | 4
Z-score | -.104 (.216) | .505 (.374)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for one month after the initiation of the intervention
Description: No difference in definitions used.
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=5) | Sham (N=4)
Psychiatric Hospitalization (Psychiatric disorders) | 1 | 0 — Hospitalization likely not causally related to study participation since it was triggered by drug use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03037983/Prot_SAP_000.pdf